CLINICAL TRIAL: NCT04349150
Title: A Pilot Study of Virtual Reality Technology as an Alternative to Pharmacological Sedation During Colonoscopy
Brief Title: Virtual Reality Alternative to Pharmacological Sedation During Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Daniel C Chung, Daniel C Chung, MD, Director of High-Risk GI Cancer Clinic, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018P001618
Record Dates: First submitted 2020-02-18; First posted 2020-04-16 (Actual); Results first posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-11

CONDITIONS: Colonoscopy
Keywords: Virtual reality

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality (Experimental): Participants on this arm will have their colonoscopy initiated under virtual reality instead of standard sedatives and narcotics
  Interventions: Device: Virtual reality

INTERVENTIONS:
Device: Virtual reality — Intervention consists of providing virtual reality in place of standard sedatives and narcotics for a portion or the duration of the colonoscopy

SUMMARY:
Colonoscopy patients will be fitted with a virtual reality head-mounted display, and virtual experiences will be initiated prior to colonoscope insertion. Colonoscopy will be initiated without standard sedatives and narcotics. The colonoscopy will proceed with the subject using virtual reality distraction instead of pharmacological sedation for as long as s/he would like. Standard sedatives and narcotics will be administered upon participant request at any time during the procedure. Questionnaires will be administered to the subject and the endoscopist after each procedure to assess the acceptability of use of virtual reality in the colonoscopy setting.

DETAILED DESCRIPTION:
This study aims to assess whether virtual reality is an acceptable alternative to pharmacological sedation during colonoscopy. Past research has shown that in order to fully experience pain, one must pay attention to it. Virtual reality has been shown to help mitigate pain by providing distraction from the painful stimulus.

In this study, participants undergo screening or surveillance colonoscopy under virtual reality distraction.

Individuals who are scheduled for a routine screening or surveillance colonoscopy and have had at least one prior colonoscopy under conscious sedation are eligible to participate. Those who give written, informed consent are fitted with and oriented to a virtual reality head-mounted display. The subject is then prepped for the colonoscopy by a registered nurse per institution protocol. This includes placement of an intravenous line.

Written consent is obtained for colonoscopy with medication by the performing endoscopist. The patient is again fitted with the virtual reality head-mounted display and virtual experiences are initiated. The endoscopist performs the colonoscopy with the subject using virtual reality distraction instead of pharmacological sedation for as long as the subject likes. Standard sedatives and narcotics will be administered by a registered nurse upon participant request at any time during the procedure.

Following the procedure, participants and endoscopists complete a questionnaire about their subjective experience with virtual reality during colonoscopy. The research coordinator fills out a case report form for each subject with information about the procedure including length, colonoscopy findings, and complications as noted by the endoscopist.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or older)
* Scheduled for screening or surveillance colonoscopy
* Has undergone at least 1 prior colonoscopy under conscious sedation

Exclusion Criteria:

* Children (<18 years)
* Scheduled to undergo colonoscopy under general anesthesia
* Scheduled to undergo colonoscopy with no sedation
* First-time colonoscopy patients
* Scheduled for colonoscopy to assess symptoms or pre-existing disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Chung, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All individuals scheduled for screening/surveillance colonoscopy who had previously undergone more than one colonoscopy under conscious sedation and were patients of any of four endoscopists at our institution were invited to participate.
Period: Overall Study
Arm/Group | Virtual Reality
Started | 31
Completed | 27
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Virtual Reality
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 1
Medical history potentially impacting exam difficulty [Count of Participants; unit: Participants]
  Abdominal/pelvic surgery | 11
  Tortuous colon | 1
  None | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Complete Colonoscopy Using Virtual Reality and no Pharmacological Rescue
Description: Measured as (x/n) * 100, where x = number of participants who completed colonoscopy using virtual reality and no pharmacological rescue, and n = total number of participants who initiated colonoscopy using virtual reality.
Time Frame: This data will be collected within 60 minutes of completion of the colonoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality
Number analyzed (Participants) | 27
Participants | 26

2. Primary Outcome: Number of Participants With Cecal Intubation
Description: Number of Participants with Cecal Intubation using virtual reality and no pharmacological sedation. Measured as x/n, where x = number of participants in whom cecal intubation is achieved when participant is using virtual reality and no pharmacological sedation, and n = total number of participants who initiated colonoscopy using virtual reality.
Time Frame: This data will be collected within 60 minutes of completion of the colonoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality
Number analyzed (Participants) | 27
Participants | 27

3. Secondary Outcome: Participant-reported Pain and Discomfort Levels
Description: participants will rate their pain and discomfort on a numeric rating scale of 1-10 (1 = no pain/discomfort, 10 = extreme pain/discomfort)
Time Frame: This data will be collected within 60 minutes of completion of the colonoscopy
Population: The 26 participants who did not request medication during colonoscopy.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Reality
Number analyzed (Participants) | 26
units on a scale
  Pain | 3.6 (1.6)
  Discomfort | 4.0 (1.4)

4. Secondary Outcome: Participant Satisfaction
Description: Participants will rate their satisfaction with their experience using virtual reality during colonoscopy on a numeric rating scale of 1-10 (1 = not satisfied, 10 = extremely satisfied).
Time Frame: This data will be collected within 60 minutes of completion of the colonoscopy
Population: The 26 participants who did not request medication during colonoscopy.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Reality
Number analyzed (Participants) | 26
units on a scale | 7.3 (2.5)

5. Secondary Outcome: Number of Participants Who Would Undergo Future Colonoscopies Using Virtual Reality and no Pharmacological Sedation
Description: Participants will rate their willingness to undergo future colonoscopies using virtual reality and no pharmacological sedation as "Yes," "Maybe," or "No."
Time Frame: This data will be collected within 60 minutes of completion of the colonoscopy
Population: The 26 participants who did not request medication during colonoscopy.
Measure: Number; unit: participants
Arm/Group | Virtual Reality
Number analyzed (Participants) | 26
participants
  Yes | 18
  Maybe | 7
  No | 1

6. Secondary Outcome: Endoscopist Satisfaction
Description: Endoscopists will rate their satisfaction performing colonoscopy on participants using virtual reality instead of pharmacological sedation on a numeric rating scale of 1-10 (1 = not satisfied, 10 = extremely satisfied).
Time Frame: This data will be collected within 60 minutes of completion of the colonoscopy
Population: The 26 participants who did not request medication during colonoscopy.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Reality
Number analyzed (Participants) | 26
units on a scale | 8.6 (1.8)

7. Secondary Outcome: Number of Endoscopies Following Which Endoscopists Indicated Willingness to Incorporate Virtual Reality Into Regular Colonoscopy Practice
Description: Endoscopists will indicate whether they would incorporate virtual reality into their regular colonoscopy practice by selecting one of the following:
  * yes
  * no
  * yes, but I would use virtual reality as an adjunct therapy rather than a standalone therapy
Time Frame: This data will be collected within 60 minutes of completion of the colonoscopy
Population: The four endoscopists participating in the study
Measure: Number; unit: Endoscopies
Arm/Group | Virtual Reality
Number analyzed (Participants) | 4
Endoscopies
  Yes | 19
  No | 0
  Yes, but I would use virtual reality as an adjunct therapy rather than a standalone therapy | 6

ADVERSE EVENTS:
Time Frame: 9 months
Description: There were no adverse events.
Arm/Group | Virtual Reality
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT04349150/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT04349150/SAP_001.pdf